CLINICAL TRIAL: NCT05787951
Title: Frequency and Risk Factors of Acute Myeloid Leukemia at Clinical Haemtology Unit of Assiut University Hospital
Brief Title: Frequency and Risk Factors of Acute Myeloid Leukemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sanaa Ezzat Hussien, Sanaa Ezzat Hussien, Assiut University
Other Study IDs: Risk factors of AML
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid | interventions — Diagnosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Bone marrow aspirite for diagnosis — Routine investigation of acute myeloid leukemia such as bone marrow aspirite for diagnosis ,cbc

SUMMARY:
1. to assess the frequency of acute myeloid leukemia at clinical Haematology unit of Assiute university hospital
2. to study correlations of known risk factors and if there are new risk factors participate in increasing frequency of acute myeloid leukemia

DETAILED DESCRIPTION:
Acute myeloid leukaemia (AML) is a rare heterogeneous disease comprising a group of hematopoietic neoplasms originating from the excessive clonal proliferation of myeloid pre- cursor cells [1]. Diagnosis of AML is based on morphological diagnosis with proliferation of blast cells ≥ 20% of bone marrow cells, flow cytometric analysis and cytogenetic abnormalities, including the t(8;21)(q22;q22), t(15;17) (q22;q12) and inv (16)(p13.1;q22) which are associated with longer remission and survival, while alterations of chromosomes 5, 7, complex karyotype and 11q23 are associated with poor response to therapy and shorter overall survival [2] The etiological agent and pathogenesis of AML are not entirely clear, only few AML cases can be accurately classified through traditional cellular morphological classification [3]It is the most common acute leukaemia in adults. It accounts for 1.3% of new cancer patients in the United States, in 2018[ 4] Some factors are well documented to increase the risk of some types of leukemia such as benzene exposure and ionizing radiation [5] increased frequency of acute myeloid leukemia has been noticed at Haematology unit so the aim of the study to assess the the frequency of acute myeloid leukemia and to evaluate the risk factors for it .

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients(above 18 years) diagnosed as acute myeloid leukemia according to WHO diagnostic criteria

Exclusion Criteria:

* Patients with other types of leukemia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Patients(above 18 years) diagnosed as acute myeloid leukemia according to WHO diagnostic criteria
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of acute myeloid leukemia at clinical Haemtology unit of Assiute university hospital | Two years

SECONDARY OUTCOMES:
Risk factors of acute myeloid leukemia at clinical Haemtology unit of Assiute university hospital | Two years

REFERENCES:
- [Background] Hwang SM. Classification of acute myeloid leukemia. Blood Res. 2020 Jul 31;55(S1):S1-S4. doi: 10.5045/br.2020.S001. PMID 32719169